CLINICAL TRIAL: NCT07338266
Title: A Single Ascending Dose Study to Assess the Safety and Pharmacokinetics of Intra-articular AVD275 Injection in Patients With Osteoarthritis of the Knee
Brief Title: Study to Assess the Safety and Pharmacokinetics of AVD275 Injection in Patients With Osteoarthritis of the Knee
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Avidence Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVD275CLIN-2025-001
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose Arm (Experimental): One low dose of AVD275 is injected to the osteoarthritic knee joint
  Interventions: Drug: AVD275 Intra-articular Injection
- Middle Dose Arm (Experimental): One middle dose of AVD275 is injected to the osteoarthritic knee joint
  Interventions: Drug: AVD275 Intra-articular Injection
- High Dose Arm (Experimental): One high dose of AVD275 is injected to the osteoarthritic knee joint
  Interventions: Drug: AVD275 Intra-articular Injection

INTERVENTIONS:
Drug: AVD275 Intra-articular Injection — A long-acting formulation of celecoxib

SUMMARY:
This study aims to understand the safety, drug concentration and distribution of an intra-articular injectable formulation of celecoxib, AVD275, in patients with knee osteoarthritis. One single injection at three different doses of the drug will be studied in a sequential order, and each participant will be monitored for 24 weeks over ten clinical visits.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate in the study; Willingness and ability to comply with the study procedures, visit schedules and follow verbal and written instructions
2. Male or female: 20 years to 75 years of age
3. Symptoms associated with OA of the knee for ≥6 months prior to screening (patient reported is acceptable); Knee OA may be unilateral or bilateral
4. Currently meets ACR Criteria (clinical and radiological) for OA as follows:

   * Knee pain
   * At least one of the following:

     1. Age > 50 years
     2. Stiffness < 30 minutes
     3. Crepitus
   * Osteophytes
5. Kellgren-Lawrence (K-L) Grade 1-4 in the index knee based on X-ray performed during screening (locally read) within 6 months from screening
6. Body mass index (BMI) ≤ 40 kg/m2
7. Ambulatory and in good general health

Exclusion Criteria:

1. Any condition that could confound the patient's assessment of index knee pain in judgement of the investigator (for example, peri-articular pain of any cause or secondary arthritis that involves the index knee, joint dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler's syndrome, hemophilia, hemochromatosis, or neuropathic arthropathy, radicular lower back pain and hip pain that is referred to the knee that could cause misclassification); Other chronic pain anywhere in the body that confounds assessment of knee or that requires the use of celecoxib
2. Malalignment of greater than 10 degrees in the femorotibial axis of the index knee on standing; Unstable joint (such as tornanterior cruciate ligament) or traumatic knee injury to the index knee (such as meniscal root tear) within 12 months of screening
3. Fibromyalgia, Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, reactive arthritis, arthritis associated with inflammatory bowel disease, crystal disease of the index knee (e.g. gout or calcium pyrophosphate deposition disease), rapidly progressive osteoarthritis (defined as joint space narrowing > 1.2 mm/year), sarcoidosis or amyloidosis
4. Effusion at screening that likely requires joint aspiration for symptom relief from day 2 to day 83 during the study, as indicated by at least four joint drainages in the past year
5. Intra-articular corticosteroids or intra-articular nonsteroidal antiinflammatory drugs (NSAIDs) (investigational or marketed) in the index knee within 2 months of screening; Intra-articular hyaluronic acid (investigational or marketed) in the index knee within 3 months of screening; Intra-articular Zilretta within 3 months of screening
6. Intramuscular or oral corticosteroids within 1 month of screening
7. Patients who received opioids (excluding tramadol and tapentadol) within 2 weeks of screening
8. Any other investigational drug/biologic use within 3 months of screening
9. Prior diagnostic arthroscopy to the index knee within 3 months of screening; Prior arthroscopic or open surgery of the index knee (including microfracture and meniscectomy) within 6 months of screening；Prior regenerative joint procedures on the index knee, including, but not limited to, stem cells transplantation, autologous chondrocyte transplantation, or mosaicplasty within 12 months of screening; History of total or partial knee arthroplasty in the index knee
10. Planned/anticipated surgery of the index knee, any other surgery, or hospitalization during the study period
11. Known hypersensitivity to any form of NSAIDs (including celecoxib), sulfonamide-containing drugs, carboxymethyl cellulose, polysorbate 80 or lidocaine; History of severe allergic reactions
12. Active or history of malignancy within the past 3 years, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the knee, or effectively managed cervical carcinoma
13. Known active or quiescent systemic fungal, bacterial (including tuberculosis), viral or parasitic infections (including HIV, hepatitis B or C viruses), or ocular herpes simplex; Any infection requiring intravenous antibiotics within 2 months of screening or oral antibiotics within 2 weeks of screening; History of infection in the index knee within 12 months of screening; History of osteomyelitis
14. Any clinically significant laboratory parameters or ECG abnormality as judged by the investigator
15. Uncontrolled diabetes as indicated by a hemoglobin A1c of >7.5% at screening
16. History of atherosclerotic cardiovascular disease (ASCVD) defined as prior myocardial infarction, stroke (ischaemic or haemorrhagic), transient ischemic attack, coronary revascularization (e.g., PCI, CABG), peripheral artery disease, or heart failure (NYHA Class II or higher) in the past three years;

    * OR a calculated 10-year ASCVD risk ≥10% based on age, sex, race, total/HDL cholesterol, systolic blood pressure, diabetes, smoking status;
    * OR current use of dual antiplatelet therapy, chronic anticoagulation (e.g., warfarin, direct oral anticoagulants), or high-dose aspirin (>300 mg/day)
17. Abnormal liver function with AST or ALT > 2 upper limit of normal (ULN) at screening
18. Abnormal kidney function with eGFR < 45 mL/min/1.73m2 at screening
19. Platelet count outside normal range at screening
20. WBC count < 3500 cells/mm3 or >20000 cells/mm3 at screening
21. Active uncontrolled psychiatric disorder including psychosis (e.g. schizophrenia), bipolar disorder, uncontrolled anxiety disorder and major depressive disorder
22. Positive drug screen (opiates, amphetamines, cocaine metabolites, benzodiazepines, cannabinoids); Active substance abuse (drugs or alcohol), history of chronic substance abuse within the past year, or prior chronic substance abuse judged by the investigator as likely to recur during the study
23. Skin breakdown at the knee where the injection would take place; Any skin condition and/or tattoo that may interfere with the evaluation of safety at the injection site
24. Women who are pregnant or nursing; Women of child-bearing potential (not surgically sterile or post-menopausal for at least 1 year as documented in medical history) not using a highly effective method of contraception (abstinence; oral, injected or implanted hormonal methods of contraception; intrauterine device or intrauterine system; condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/cream/suppository; or male sterilization (vasectomy for at least 3 months))
25. Any other clinically significant acute or chronic medical conditions (e.g. bleeding disorder) that, in the judgement of the investigator, would preclude the use of an intra-articular NSAID or that could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment emergent adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ang Li, Study Director — Avidence Therapeutics
Locations (1):
- Cognivus Research Group, Wahroonga, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided